CLINICAL TRIAL: NCT05012020
Title: Feasibility Study of a Smartphone-based Patient Application and Web-based Clinic Portal Platform for Remote Patient Monitoring of Chronic Kidney Disease and Peritoneal Dialysis Patients
Brief Title: Feasibility Study of a mHealth Platform for Remote Patient Monitoring of CKD and Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AWAK Technologies Pte Ltd (Industry)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SG-CLI-DOC-328
Record Dates: First submitted 2021-07-22; First posted 2021-08-19 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Digital Health; mHealth; Remote patient monitoring; Chronic care management
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mHealth Remote Monitoring (Experimental): Use of the Clinic Portal by Healthcare professionals and use of the Mobile App by patients/caregivers
  Interventions: Device: mHealth Remote Monitoring platform

INTERVENTIONS:
Device: mHealth Remote Monitoring platform — Clinic Portal and Mobile Application for remote monitoring of Chronic Kidney Disease patients and patients on Peritoneal Dialysis

SUMMARY:
The best treatment of Chronic Kidney Disease (CKD) is facilitated by early detection, when the progression of the disease can be slowed down or stopped. Early treatment focuses on diet, exercise, lifestyle changes, treating risk factors (diabetes, hypertension, etc.) and administration of medications supporting kidney functions. However, once the glomerular filtration rate dropped below 15 ml/min/1.73m2, treatment with dialysis or a kidney transplant is required. Dialysis treatments come with a huge lifestyle management and economic burden to the patients as well as the healthcare systems.

The challenges may be facilitated by usage of mobile applications that help the patients/caregivers and multidisciplinary team to manage the complexity of Peritoneal Dialysis (PD) treatment. Even though several mobile applications currently exist, they focus on certain limited aspects of health monitoring like diet or vitals and medical adherence like medication reminders. An application which would take a comprehensive all-in-one solution approach targeted towards managing kidney health is needed. The platform developed by AWAK Technologies consists of a Admin Portal, web-based Clinic Portal and a Patient Mobile Application. The App would allow patients/caregivers to enter treatment data related to their dialysis therapy, medication, symptoms and vital monitoring. It also allows them to communicate with their healthcare team via messaging and teleconsult.

The study aims to evaluate the feasibility of using this mHealth platform in the clinical setting. Additionally, the clinical investigation seeks to obtain data for further development of the mHealth platform that will better fulfil the needs of patients and healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CKD or on PD
* Treated at the Singapore General Hospital's Renal Clinic
* Able to read and understand English language well enough to independently follow instructions in the App and enter data in English
* Cognitively and physically capable and willing to interact with a digital device with internet access and perform self measurements
* Owns a digital device with internet access [Apple/Android running on at least iPhone operating system (iOS) v13/Android v9]

Exclusion Criteria:

* Living in an assisted facility, e.g., eldercare facilities, and hospices where their care is done/provided completely by healthcare professionals
* Patients or caregivers who have no access to digital device with internet access
* Patient has a severe comorbidity or poor general physical/mental health that, in the opinion of the investigator, will not allow the patient to be a good investigation candidate (i.e., other disease processes, mental capacity, substance abuse, shortened life expectancy, vulnerable patient population)
* The patient is currently involved in another clinical investigation where that participation may conflict or interfere with the treatment, follow-up or results of this clinical investigation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adherence to mobile app use as assessed by total number of participants adhering to mobile app use out of all participants. | 6 months
  Adherence is defined as use of app for ≥ 2 times on average per week for CKD patients and 7 times on average per week for PD patients
Average time spent on using mobile app per day per participant | 6 months
  Reported as minutes per day per participant

SECONDARY OUTCOMES:
Frequency of smart companion devices use | 6 months
  Assessed by average number of smart device use per week per participant (reported as frequency per week per participant)
User experience | 6 months
  Measured by the mHealth app usability questionnaire (7-point likert scale with total possible score of 147)
Pre and post study comparison of hospitalization rate | 6 months
  Reported as days per patient-month
Pre and post study comparison of total number of unplanned clinic visit or emergency department visit | 6 months
Pre and post study comparison of exit-site infection rate among peritoneal dialysis patients | 6 months
  Reported as episode per patient-year
Pre and post study comparison of peritonitis rate for PD patients | 6 months
  Reported as episode per patient-year
Pre and Post study comparison of estimated Glomerular Filtration Rate (eGFR) for CKD patients | 6 months
Pre and Post study comparison of blood pressure measurement for CKD patients | 6 months
Pre and Post study comparison of the number of anti-hypertensive medications for CKD patients | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Htay Htay, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore